CLINICAL TRIAL: NCT02114554
Title: Clinical Characteristics and Prognostic Factors of Mitochondrial nt3243 A>G Mutation in Taiwan
Brief Title: Mitochondrial nt3243 A>G Mutation in Taiwan
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201307058RINB
Record Dates: First submitted 2014-02-09; First posted 2014-04-15 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: MELAS Syndrome; Noninsulin-dependent Diabetes Mellitus With Deafness
Keywords: MELAS; MIDD; Heteroplasmy
MeSH Terms: conditions — MELAS Syndrome; Noninsulin-dependent diabetes mellitus with deafness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Mitochondrial diseases are multisystem disorders that present with a wide range of clinical manifestations. Mitochondrial DNA nt3243A>G mutation is one of the most common mutations seen in mitochondrial diseases. Syndromes associated with this mutation include mitochondrial encephalopathy, lactic acidosis, and stroke-like episodes (MELAS), maternally inherited diabetes and deafness (MIDD), myoclonic epilepsy with ragged red fibers (MERRF), and chronic progressive external ophthalmoplegia (CPEO). Clinical analyses of mitochondrial DNA nt3243A>G mutation from Taiwan remain scarce. The present study aims to investigate the clinical features and prognostic factors of patients with mt3243A>G mutation in Taiwan.

DETAILED DESCRIPTION:
Patients and clinical features. The study will be carried out at National Taiwan University hospital, a tertiary medical center in Taipei. The Medical Genetics Department at National Taiwan University Hospital receives referral and conducts genetic testing for hospitals all around Taiwan. We will review the medical chart of all patients with documented mitochondrial DNA nt3243 point mutation. Demographic data, age at onset of symptoms, clinical features (including stroke, seizure-like episode, lactic level, diabetes mellitus, hearing impairment, myopathy, electrocardiogram abnormality, chronic progressive external ophthalmoplegia), relevant family history, treatment, and outcome will be recorded. Full MELAS phenotype was defined as the presence of focal central nervous system events, either seizures, strokes, or both.

Genetic analysis. Genomic DNA was extracted from peripheral blood leukocytes using the Puregene DNA purification kit (Gentra Systems, Minneapolis, Minnesota, USA). Polymerase chain reaction (PCR) for mitochondrial DNA nt3243 point mutation was carried out by left primer 5'-cggagtaatccaggtcggtt-3' and right primer 5'-ggaattgaacctctgactgt-3'. Presence of mitochondrial DNA nt3243 A>G mutation was detected after Hae III restriction enzyme digestion.

Heteroplasmy of mitochondrial nt3243A>G mutation was detected by real-time amplification refractory mutation system quantitative PCR (ARMS-qPCR) assay as previously reported [19]. In brief, wild-type and mutant-target primers, each 500 nM, were added into a 10-ml PCR reaction containing 1X KAPA SYBR® FAST ABI Prism® qPCR Master Mix (KAPABIOSYSTEMS, Cat No. KK4603) and 4 ng of genomic DNA. Real-time PCR conditions were 2 min at 50°C, 20 seconds at 95°C, followed by 40 cycles of 15 seconds of denaturation at 95°C and 30 seconds of annealing/extension at 62°C. Data of cross point and concentration fluorescent signal intensity of PCR products was recorded and analyzed by ABI StepOnePlusTM Real-Time PCR System (Applied Biosystems) and StepOne software v2.1 (Applied Biosystems). The threshold cycle ( CT value) within the linear exponential phase was used to construct the standard curve and to measure the original copy number of DNA template. The percentage of the mutant mtDNA was calculated using formula as below: Heteroplasmy %= 1/(1+ 1/2△CT).

Statistical analysis. SPSS 17.0 (SPSS, Chicago, IL, USA) was used for statistical analysis. Results were given as median and range, or mean ± 1 SD, when appropriate. Student 's t-test was used to compare unpaired groups. Fisher's exact test was used to determine associations between two categorical variables. Cox-regression model was used to analyze possible prognostic factors. Inter-group differences at outcome were compared by Kaplan-Meier estimate and log-rank test. Pearson's correlation was used to correlate heteroplasmy to age of diagnosis. A p value < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

-Patients with mitochondrial DNA nt3243 A>G mutation

Exclusion Criteria:

-Patients without confirmed mitochondrial DNA nt3243 A>G mutation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with mitochondrial DNA nt3243 A>G mutation detected at National Taiwan University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Prognostic factors for poor outcome | Within follow-up period, which is estimated to be 5 years in average.
  Poor outcome includes death and development of poor performance (a modified Rankin scale 4 or higher). Univariate and multivariate analyses will be utilized to study whether specific clinical presentations (for instance, the presence of stroke, seizure, diabetes, etc.) and degree of heteroplasmy are associated with poor outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Lin Lee, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan